CLINICAL TRIAL: NCT05949489
Title: Associations Between Psychological Factors, Pain Sensitivity, and Physical Function in Knee Osteoarthritis: a One-year Follow up Study
Brief Title: Psychological and Pain Factors in Knee Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: Knee OA Study 01
Record Dates: First submitted 2023-07-07; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Knee Osteoarthritis: Patients with physician-diagnosed knee osteoarthritis
  Interventions: Diagnostic Test: WOMAC pain subscale

INTERVENTIONS:
Diagnostic Test: WOMAC pain subscale — The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale is a self-reported questionnaire that is used to measure pain in people with osteoarthritis (OA). The subscale consists of five items that ask about the intensity, frequency, and duration of pain in the hip and knee joints.
  The WOMAC Pain Subscale has been shown to be a reliable and valid measure of pain in people with OA. It has been used in a number of clinical trials and is considered to be a standard measure of pain in OA.
  The WOMAC Pain Subscale is scored on a scale of 0 to 4, with 0 indicating no pain and 4 indicating severe pain. The total score for the subscale is the sum of the scores for the five items. A higher score indicates more pain.

SUMMARY:
This study aims to determine if baseline measures of psychology and pain sensitivity can predict changes in physical function at 1 year in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of knee OA based on clinical and radiographic ACR criteria
* Pain in or around the knee on most days of the past month
* Aged 40 years or above
* Ambulatory with or without walking aid

Exclusion Criteria:

* Inflammatory arthritis (rheumatoid arthritis, lupus, etc.)
* Recent knee injury or surgery (past 3 months)
* Severe comorbidity likely to prevent study completion (dementia, terminal illness)
* inability to comply with study procedures or follow up

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical knee osteoarthritis experiencing persistent knee pain.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Function from Baseline to 1 year (WOMAC) | Change from baseline at 1 year
  Assessed using the WOMAC physical function subscale (0-68 scale, higher = worse function)

SECONDARY OUTCOMES:
Pain Catastrophizing Scale | Change from baseline at 1 year
  Assessed using the Pain Catastrophizing Scale (0-52 scale, higher = higher catastrophizing)
Kinesiophobia | Change from baseline at 1 year
  Assessed using the Tampa Scale of Kinesiophobia (17-68 scale, higher = higher kinesiophobia)
Change in Sleep Quality from Baseline to 1 year (Pittsburgh Sleep Quality Index) | Change from baseline at 1 year
  Assessed using the Pittsburgh Sleep Quality Index (0-21 scale, higher = worse sleep quality)
Change in Pain Self-efficacy from Baseline to 1 year (Pain Self-Efficacy Questionnaire) | Change from baseline at 1 year
  Assessed using the Pain Self-Efficacy Questionnaire (0-60 scale, higher = stronger self-efficacy beliefs)

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No